CLINICAL TRIAL: NCT02009163
Title: A Phase 3, Multicenter, Double-blind, Placebo-controlled, Randomized-withdrawal Study to Evaluate the Maintenance of Efficacy of SPD489 in Adults Aged 18-55 Years With Moderate to Severe Binge Eating Disorder
Brief Title: Evaluate the Maintenance of Efficacy of SPD489 in Adults Aged 18-55 Years With Moderate to Severe Binge Eating Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-346; 2012-004457-88 (EudraCT Number)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine dimesylate (Experimental): Administer one capsule (50 or 70 mg) orally daily at approximately 7:00 AM.
  Interventions: Drug: Lisdexamfetamine dimesylate
- Placebo (Placebo Comparator): Administer one capsule orally daily at approximately 7:00 AM.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — SDP489 30, 50, or 70mg capsule once per day (open-label and double-blind periods)
  Other Names: SPD489; LDX
  Arms: Lisdexamfetamine dimesylate
Other: Placebo — Placebo capsule once per day (double-blind period)
  Arms: Placebo

SUMMARY:
To evaluate maintenance of efficacy based on time to relapse between SPD489 (50 or 70mg) and placebo, as measured by the number of binge days (defined as days during which at least 1 binge episode occurs) per week as assessed by clinical interview based on subject diary and Clinical Global Impression - Severity (CGI-S) scores for patients who responded to SPD489 by the end of the Open-label Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18-55 years of age, inclusive.
2. Subject meets the following criteria for a diagnosis of BED:

   * Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following: eating, in a discrete period of time (eg, within a 2-hour period) an amount of food that is definitely larger than most people would eat in a similar period of time under similar conditions, and a sense of lack of control over the eating (eg, a feeling that one cannot stop eating or control what or how much one is eating).
   * The binge eating episodes are associated with at least 3 of the following: eating much more rapidly than normal; eating until uncomfortably full; eating large amounts of food when not feeling physically hungry; eating alone because of being embarrassed by how much one is eating; feeling disgusted with oneself, depressed, or feeling very guilty after overeating.
   * Marked distress regarding binge eating.
   * The binge eating occurs, on average, at least 2 days a week for 6 months.
   * The episodes of binge eating do not occur exclusively during the course of bulimia nervosa or anorexia nervosa.
3. Subject is consistently able to swallow a capsule.

Exclusion Criteria:

1. Subject has current diagnosis of bulimia nervosa or anorexia nervosa.
2. Subject is receiving psychotherapy or weight loss support within the past 3 months.
3. Subject has used psychostimulants to facilitate fasting or dieting within the past 6 months.
4. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease.
5. Subject has abnormal thyroid function.
6. Subject initiated treatment with a lipid lowering medication within the past 3 months.
7. Subject has a history of moderate or severe hypertension.
8. Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder.
9. Subject has glaucoma.
10. Subject is female and pregnant or nursing.
11. Subjects who have had bariatric surgery, lap bands, duodenal stents, or other procedures for weight loss.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 418 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2015-04-08 (Actual); Study Completion 2015-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (53):
- United States (39):
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - Compass Research LLC North Clinic, Leesburg, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Scientific Clinical Research, Inc, North Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - NeuroTrials Research, Inc, Atlanta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - Cypress Medical Research Center, Wichita, Kansas
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - McLean Hospital, Belmont, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - HBSA-Pacific Institute for Research & Evaluation, Albuquerque, New Mexico
  - Brooklyn Medical Institute, Brooklyn, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Linder Center of Hope, Mason, Ohio
  - Oregon Center for Clinical Investigations, Inc (OCCI, Inc), Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc (OCCI, Inc), Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Inc, Anderson, South Carolina
  - Radiant Research, Inc, Greer, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solution, Inc, Memphis, Tennessee
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Texas Center for Drug Development, Inc, Houston, Texas
  - Research Across America, Plano, Texas
  - Radiant Research, Inc, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
- Canada (2):
  - Anxiety and Mood Disorder Center, Mississauga, Ontario
  - Manna Research, Pointe-Claire, Quebec
- Germany (6):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - EMOVIS GmbH - Klinische Forschung, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Forschung Schwerin GmbH, Friedrichstrasse 1, Schwerin
  - Studienzentrum Nordwest, Westerstede
- Spain (3):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital del Henares, Madrid
- Sweden (3):
  - Lakarmottagningen Ekdahl & Kronberg, Malmo
  - Sofiahemmet, Stockholm
  - Stockholm Center for Eating Disorders, Stockholm

REFERENCES:
- [Derived] Robertson B, Wu J, Fant RV, Schnoll SH, McElroy SL. Assessment of Amphetamine Withdrawal Symptoms of Lisdexamfetamine Dimesylate Treatment for Adults With Binge-Eating Disorder. Prim Care Companion CNS Disord. 2020 Mar 26;22(2):19m02540. doi: 10.4088/PCC.19m02540. PMID 32237290
- [Derived] Hudson JI, McElroy SL, Ferreira-Cornwell MC, Radewonuk J, Gasior M. Efficacy of Lisdexamfetamine in Adults With Moderate to Severe Binge-Eating Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):903-910. doi: 10.1001/jamapsychiatry.2017.1889. PMID 28700805

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD489 (Open-label Period): SPD489 treatment was taken orally once daily at approximately 7:00 AM. All participants began treatment with SPD489 at the lowest dose level (30mg) during the 4-week open-label dose-optimization period. After 1 week of treatment at 30mg, all participants were titrated to the next dose level (50mg). After 1 week of treatment at 50mg, all participants were titrated to the highest dose level (70mg), as tolerated and as clinically indicated. After 1 week of treatment at the highest dose, the participant could have been down-titrated to 50mg; no further dose adjustments were permitted. The optimal daily dose of 50 or 70mg achieved during dose-optimization was maintained throughout the 8-week dose-maintenance period. The total time of the open-label period was 12 weeks.
- Placebo (Randomized-withdrawal Period): During the 26-week double-blind randomized-withdrawal phase, participants randomized to placebo received matching placebo capsules daily. After the 26-week double-blind randomized-withdrawal phase, participants were followed for 1 week.
- SPD489 (Randomized-withdrawal Period): For participants randomized to SPD489, the optimal daily dose of 50 or 70mg was continued throughout the 26-week double-blind randomized-withdrawal phase. After the 26-week double-blind randomized-withdrawal phase, participants were followed for 1 week.
Period: Open-label Period (Non-randomized)
Arm/Group | SPD489 (Open-label Period) | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Started | 418 | 0 | 0
Completed | 275 | 0 | 0
Not Completed | 143 | 0 | 0
Not completed — Failure to Meet Randomization Criteria | 48 | 0 | 0
Not completed — Withdrawal by Subject | 29 | 0 | 0
Not completed — Adverse Event | 22 | 0 | 0
Not completed — Lost to Follow-up | 20 | 0 | 0
Not completed — Protocol Violation | 10 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Other | 13 | 0 | 0
Period: Randomized-withdrawal Period
Arm/Group | SPD489 (Open-label Period) | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Started | 0 (The open-label treatment group is not an arm of the randomized-withdrawal period.) | 138 (The total who started the Placebo and SPD489 arms equals those who completed the open-label period.) | 137 (The total who started the Placebo and SPD489 arms equals those who completed the open-label period.)
Completed | 0 | 50 | 102
Not Completed | 0 | 88 | 35
Not completed — Withdrawal by Subject | 0 | 25 | 9
Not completed — Lost to Follow-up | 0 | 13 | 6
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Relapse Criteria Met | 0 | 40 | 5
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Other | 0 | 9 | 5

BASELINE CHARACTERISTICS:
Population: The Open-label Safety Population (OSP) was defined as all participants who had taken at least 1 dose of SPD489 in the open-label period and who had a post-baseline safety assessment. Seven participants were enrolled but not treated and thus not included in the OSP.
Groups:
- Open-label Safety Population: The Open-label Safety Population included all participants who had taken at least 1 dose of SPD489 in the open-label period and who had a post-baseline safety assessment.
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.40)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years of age | 217
  >/= 40 years of age | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse From Date of Randomization to Endpoint of The Randomized-withdrawal Period
Description: Relapse status was assessed during the double-blind treatment phase and was defined as having 2 or more binge days per week for 2 consecutive weeks (14 consecutive days) prior to any visit and having an increase in Clinical Global Impressions-Severity (CGI-S) score of 2 or more points compared to the randomized-withdrawal baseline (date of relapse - date of randomization). Binge eating information was captured via a self-report paper diary. The binge diary captured the number of binges per day, total hours per day spent binging, type of binge (at mealtime or at another time other than mealtime), and a description of the binge (amounts and types of foods). Binge frequency was reviewed by the clinician with the subject to confirm reported binge episodes per day. The CGI-S was performed to rate the severity of a subject's condition using a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill).
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: The Full Analysis Set (FAS): participants in the Randomized Safety Analysis Set (RSAS) with at least 1 post-randomization CGI-S assessment. Three participants in the placebo group were randomized and included in the RSAS but not in the FAS. Visit 21 could include participants who discontinued but completed a final safety and efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 131 | 136
days | NA [55.0 to NA] — As neither treatment group had over 50% of subjects experiencing relapse during the 26-week randomized-withdrawal phase, the median time to relapse and inter-quartile range was not calculable. | NA [NA to NA] — As neither treatment group had over 50% of subjects experiencing relapse during the 26-week randomized-withdrawal phase, the median time to relapse and inter-quartile range was not calculable.
Statistical Analysis 1: Comparison: Placebo (Randomized-withdrawal Period) vs SPD489 (Randomized-withdrawal Period); Test type: Superiority or Other; p < 0.001, Log Rank — P-value based on a log-rank test, stratified by 4-week cessation status (Yes, No). 4-week cessation was defined as a subject having no binge days during the 4 weeks prior to randomization

2. Secondary Outcome: Change From Randomized-Withdrawal Baseline in The Number of Binge- Eating Days Per Week During The Randomized-withdrawal Period
Description: A binge day was defined as days during which at least 1 binge episode occurred. As assessed by clinical interview based on subject binge diary. Binge eating information was captured via a self-report paper diary. The binge diary captured the number of binges per day, total hours per day spent binging, type of binge (at mealtime or at another time other than mealtime), and a description of the binge (amounts and types of foods). Binge frequency was reviewed by the clinician with the subject to confirm reported binge episodes per day. A negative change from Baseline indicates that binge-related behavior decreased. The randomized -withdrawal-baseline was defined as the weekly average number of binge days for the 14 days prior to the Randomization Visit (Visit 8).
Time Frame: Randomized--withdrawal baseline (Visit 8; 12 weeks after start of open- label treatment [Week 12]), Visit 21 (26 weeks after randomization [Week 38])
Population: The FAS. Three participants in the placebo group were randomized and included in the RSAS but not in the FAS. Not all participants in the FAS had data collected for this outcome. Visit 21 included only participants who completed randomized treatment (placebo: n=50; SPD489: n=102).
Measure: Least Squares Mean (Standard Error); unit: days
Groups:
- SPD489 (Randomized--Withdrawal Period): For participants randomized to SPD489, the optimal daily dose of 50 or 70 mg was continued throughout the 26-week double-blind randomized--withdrawal phase. After the 26-week double-blind randomized-withdrawal phase, participants were followed for 1 week.
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized--Withdrawal Period)
Number analyzed (Participants) | 131 | 136
days | 0.63 (0.076) | 0.02 (0.061)
Statistical Analysis 1: Comparison: Placebo (Randomized-withdrawal Period) vs SPD489 (Randomized--Withdrawal Period); Test type: Superiority or Other; p < 0.001, mixed- effects model for repeated measur — Nominal P-value not adjusted for multiplicity; MMRM over all post-randomization visits during the randomized-withdrawal phase. Value for change from baseline = outcome variable; difference in LS mean = -0.61, 95% CI 2-sided [-0.81 to -0.42]

3. Secondary Outcome: Percent of Participants Within Each Category of The Clinical Global Impression-Severity of Illness (CGI-S) Scale at Endpoint of The Randomized-withdrawal Period
Description: The CGI-S permits a global evaluation of a subject's condition and severity of symptoms. The CGI-S was performed to rate the severity of a subject's condition based on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill).
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: The FAS. Three participants in the placebo group were randomized and included in the RSAS but not in the FAS. Visit 21 could include participants who discontinued but completed a final safety and efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 131 | 136
percentage of participants
  Normal, Not at All Ill | 45.0 | 81.6
  Borderline Mentally Ill | 10.7 | 11.8
  Mildly Ill | 14.5 | 2.2
  Moderately Ill | 22.1 | 2.2
  Markedly Ill | 6.9 | 2.2
  Severely Ill | 0.0 | 0.0
  Among the Most Extremely Ill | 0.8 | 0.0
Statistical Analysis 1: Comparison: Placebo (Randomized-withdrawal Period) vs SPD489 (Randomized-withdrawal Period); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted P-value for the difference in distribution between treatment groups in CGI-S; Cochran-Mantel-Haenszel test with a modified ridit score, adjusting for Visit 8 (Week 12) CGI-S as the covariate

4. Secondary Outcome: Change From Randomized-Withdrawal Baseline in The Total Score of The Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) During The Randomized-withdrawal Period
Description: The Y-BOCS-BE measures the obsession of binge eating thoughts and compulsiveness of binge eating behaviors. The scale is a clinician rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms). The scale includes questions regarding the amount of time spent on obsessions, impairment or distress experienced, and resistance and control over these thoughts. The same types of questions were asked about compulsions (ie, time spent, interference, etc.).Total scores range from 0 to 40. A total score of 0-7 is sub-clinical, 8-15 is mild, 16-23 is moderate, 24-31 is severe, and 32-40 is extreme. A decrease from baseline in Y-BOCS-BE Total Score represents an improvement in obsession with binge-eating thoughts or compulsiveness of binge-eating behaviors.
Time Frame: Randomized-withdrawal baseline (Visit 8; 12 weeks after start of open-label treatment [Week 12]), Visit 21 (26 weeks after randomization [Week 38])
Population: The FAS. Three participants in the placebo group were randomized and included in the RSAS but not in the FAS. Not all participants in the FAS had data collected for this outcome. Visit 21 included only participants who completed randomized treatment (placebo: n=54; SPD489: n=107).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 131 | 136
units on a scale | 5.5 (0.66) | -0.0 (0.52)
Statistical Analysis 1: Comparison: Placebo (Randomized-withdrawal Period) vs SPD489 (Randomized-withdrawal Period); Test type: Superiority or Other; p < 0.001, mixed-effects model for repeated measure — Nominal P-value not adjusted for multiplicity; [statistical method as in outcome 2, analysis 1]; difference in LS mean = -5.6, 95% CI 2-sided [-7.2 to -3.9]

5. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Mobility at Endpoint of The Open-label Period
Description: The EuroQoL Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) is a health-related quality of life (QoL) measure that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression as well as current overall health. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses, from poor health to good health.
Time Frame: Visit 8 (12 weeks after start of open-label treatment [Week 12] or Early Termination)
Population: The Open-label Safety Population (OSP), defined as participants who had taken at least 1 dose of SPD489 in the open-label period and who had a post-baseline safety assessment. Not all participants had data collected for this outcome. Visit 8 could include participants who discontinued but completed a safety and efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 397
percentage of participants
  I have no problems in walking about | 87.9
  I have slight problems in walking about | 9.8
  Moderate problems in walking about | 1.5
  I have severe problems in walking about | 0.8
  I am unable to walk about | 0

6. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5--Dimension 5--Level Self--Report Questionnaire (EQ--5D--5L) For Mobility at Endpoint of The Randomized-withdrawal Period
Description: as for outcome 5
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: The FAS. Three participants in the placebo group were randomized and included in the RSAS but not in the FAS. Not all participants in the FAS had data collected for this outcome. Visit 21 could include participants who discontinued but completed a final safety and efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 116 | 127
percentage of participants
  I have no problems in walking about | 83.6 | 91.3
  I have slight problems in walking about | 14.7 | 6.3
  Moderate problems in walking about | 1.7 | 1.6
  I have severe problems in walking about | 0.0 | 0.8
  I am unable to walk about | 0.0 | 0.0

7. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Self Care at Endpoint of The Open-label Period
Description: as for outcome 5
Time Frame: Visit 8 (12 weeks after start of open-label treatment [Week 12] or Early Termination)
Population: The OSP. Not all participants had data collected for this outcome. Visit 8 could include participants who discontinued but completed a safety and efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 397
percentage of participants
  I have no problems washing or dressing myself | 98.7
  I have slight problems washing or dressing myself | 0.8
  Moderate problems washing or dressing myself | 0.3
  I have severe problems washing or dressing myself | 0.3
  I am unable to wash or dress myself | 0

8. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Self Care at Endpoint of The Randomized-withdrawal Period
Description: as for outcome 5
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: The FAS. Three participants in the placebo group were randomized and included in the RSAS but not included in the FAS. Not all participants in the FAS had data collected for this outcome. Visit 21 could include participants who discontinued but completed a final safety and efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 116 | 127
percentage of participants
  I have no problems washing or dressing myself | 98.3 | 98.4
  I have slight problems washing or dressing myself | 0.9 | 0.8
  Moderate problems washing or dressing myself | 0.9 | 0.8
  I have severe problems washing or dressing myself | 0.0 | 0.0
  I am unable to wash or dress myself | 0.0 | 0.0

9. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Usual Activities at Endpoint of The Open-label Period
Description: as for outcome 5
Time Frame: Visit 8 (12 weeks after start of open-label treatment [Week 12] or Early Termination)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 397
percentage of participants
  I have no problems doing my usual activities | 88.9
  I have slight problems doing my usual activities | 8.1
  Moderate problems doing my usual activities | 2.3
  I have severe problems doing my usual activities | 0.8
  I am unable to do my usual activities | 0

10. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Usual Activities at Endpoint of The Randomized-withdrawal Period
Description: as for outcome 5
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 116 | 127
percentage of participants
  I have no problems doing my usual activities | 79.3 | 86.6
  I have slight problems doing my usual activities | 16.4 | 11.0
  Moderate problems doing my usual activities | 2.6 | 0.8
  I have severe problems doing my usual activities | 0.0 | 1.6
  I am unable to do my usual activities | 1.7 | 0.0

11. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Pain and Discomfort at Endpoint of The Open-label Period
Description: as for outcome 5
Time Frame: Visit 8 (12 weeks after start of open-label treatment [Week 12] or Early Termination)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 397
percentage of participants
  I have no pain or discomfort | 72.3
  I have slight pain or discomfort | 20.9
  Moderate pain or discomfort | 5.3
  I have severe pain or discomfort | 1.3
  I have extreme pain or discomfort | 0.3

12. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Pain and Discomfort at Endpoint of The Randomized-withdrawal Period
Description: as for outcome 5
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 116 | 127
percentage of participants
  I have no pain or discomfort | 75.0 | 71.7
  I have slight pain or discomfort | 16.4 | 18.1
  Moderate pain or discomfort | 8.6 | 8.7
  I have severe pain or discomfort | 0.0 | 0.0
  I have extreme pain or discomfort | 0.0 | 1.6

13. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Anxiety And Depression at Endpoint of The Open-label Period
Description: as for outcome 5
Time Frame: Visit 8 (12 weeks after start of open-label treatment [Week 12] or Early Termination)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 397
percentage of participants
  I am not anxious or depressed | 80.9
  I am slightly anxious or depressed | 15.6
  Moderately anxious or depressed | 2.3
  I am severely anxious or depressed | 1.0
  I am extremely anxious or depressed | 0.3

14. Secondary Outcome: Percent of Participants Within Each Category of The EuroQuol Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Anxiety And Depression at Endpoint of The Randomized-withdrawal Period
Description: as for outcome 5
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 116 | 127
percentage of participants
  I am not anxious or depressed | 66.4 | 79.5
  I am slightly anxious or depressed | 26.7 | 15.7
  Moderately anxious or depressed | 4.3 | 3.1
  I am severely anxious or depressed | 2.6 | 0.8
  I am extremely anxious or depressed | 0.0 | 0.8

15. Secondary Outcome: Number of Participants With a Positive Response on The Columbia Suicide Severity Rating Scale (C-SSRS) at Endpoint of The Open-label Period
Description: The C-SSRS is a semistructured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The interview was initiated with 5 (yes/no) questions, presented in ascending order of severity, about suicidal ideation. The most severe type of ideation was rated for frequency, duration, controllability, deterrents, and reason. If the answer to the first 2 ideation questions was "yes," the clinician asked questions 3-5. Active suicidal ideation included any participant who answered "yes" to questions 2-5. If the answers to ideation questions 1 and 2 were "No," then the clinician proceeded to 5 (yes/no) questions that addressed suicidal behavior, which was categorized as actual attempt, interrupted attempt, aborted attempt, preparatory acts or behaviors, and completed suicide.
Time Frame: Visit 8 (12 weeks after start of open-label treatment [Week 12])
Population: The OSP. Three participants in the OSP did not have data collected for this outcome. Visit 8 included only participants who completed open-label treatment.
Measure: Number; unit: participants
Groups:
- Open-label Safety Population: The Open-label Safety Population included all participants who had taken at least 1 dose of SPD489 in the open-label phase and who had a post-baseline safety assessment.
Arm/Group | Open-label Safety Population
Number analyzed (Participants) | 408
participants
  Suicidal Behavior | 0
  Active Suicidal Ideation | 0
  Non-Suicidal Self-Injurious Behavior | 2

16. Secondary Outcome: Number of Participants With a Positive Response on The Columbia Suicide Severity Rating Scale (C-SSRS) at Endpoint of The Randomized-withdrawal Period
Description: as for outcome 15
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination)
Population: The Randomized Safety Analysis Set (RSAS), defined as participants in the SAS who were randomized and took at least 1 dose of investigational product in the randomized-withdrawal period. Four (placebo) and one (SPD489) participants were randomized but not treated and thus not included in the RSAS. Three participants had no data for this outcome.
Measure: Number; unit: participants
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 131 | 136
participants
  Suicidal Behavior | 0 | 0
  Active Suicidal Ideation | 0 | 0
  Non-Suicidal Self-Injurious Behavior | 0 | 1

17. Secondary Outcome: Total Scores For The Amphetamine Cessation Symptom Assessment (ACSA) Scale During Follow-up
Description: The ACSA was used in this study to assess potential withdrawal symptoms associated with chronic use of SPD489. The ACSA is a self-completed scale used to assess withdrawal symptoms. The scale has 16 symptom items rated on a 5-point scale ranging from 0 (not at all) to 4 (extremely). The ACSA total score ranges from 0-64, where a higher score indicates greater withdrawal symptom severity.
Time Frame: Visit 21 (26 weeks after randomization [Week 38] or Early Termination) and Visit 22 (7 days post last dose)
Population: The RSAS. Four (placebo) and one (SPD489) participants were randomized but not treated and thus not included in the RSAS. Visits 21 and 22 could include participants who discontinued but completed a final safety and efficacy assessment. Not all participants had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Number analyzed (Participants) | 134 | 136
units on a scale
  Visit 21, n=88, 94 | 7.6 (8.33) | 4.9 (7.81)
  Visit 22, n=75, 78 | 4.6 (5.84) | 5.3 (7.98)

ADVERSE EVENTS:
Description: Treatment emergent AEs are reported for the Open-label Safety Population and Randomized Safety Analysis Set (Randomized-withdrawal Period). Seven participants were enrolled but not treated or included in the Open-label Safety Population. Four (placebo) and one (SPD489) participants were randomized but not treated and thus not included in the RSAS.
Groups:
- Placebo (Randomized-withdrawal Period): During the 26-week double-blind randomized-withdrawal phase, participants randomized to placebo received matching placebo capsules daily. After the 26-week double-blind randomized-withdrawal phase, participants were followed for 1 week .
Arm/Group | SPD489 (Open-label Period) | Placebo (Randomized-withdrawal Period) | SPD489 (Randomized-withdrawal Period)
Serious Adverse Events (participants affected / at risk) | 3/411 | 0/134 | 2/136
Other Adverse Events (participants affected / at risk) | 303/411 | 45/134 | 59/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 (Open-label Period) (N=411) | Placebo (Randomized-withdrawal Period) (N=134) | SPD489 (Randomized-withdrawal Period) (N=136)
Congenital Anomaly in Offspring (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nerve Root Compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 (Open-label Period) (N=411) | Placebo (Randomized-withdrawal Period) (N=134) | SPD489 (Randomized-withdrawal Period) (N=136)
Dry mouth (Gastrointestinal disorders) | 139 (145) | 2 (2) | 7 (7)
Headache (Nervous system disorders) | 66 (84) | 9 (9) | 12 (14)
Insomnia (Psychiatric disorders) | 46 (46) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 38 (44) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 35 (37) | 3 (3) | 6 (6)
Anxiety (Psychiatric disorders) | 29 (32) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 28 (29) | 1 (1) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 23 (24) | 0 (0) | 3 (3)
Feeling jittery (General disorders) | 21 (26) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 21 (24) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 20 (20) | 9 (9) | 13 (15)
Irritability (General disorders) | 19 (22) | 4 (5) | 4 (4)
Fatigue (General disorders) | 18 (19) | 7 (7) | 4 (4)
Tachycardia (Cardiac disorders) | 17 (20) | 0 (0) | 2 (3)
Blood pressure increased (Investigations) | 15 (17) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 14 (16) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 14 (14) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 13 (13) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 5 (7) | 11 (12)
Dizziness (Nervous system disorders) | 10 (11) | 0 (0) | 1 (4)
Thirst (General disorders) | 9 (11) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (10) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3) | 5 (5)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (4) | 4 (4)
Initial insomnia (Psychiatric disorders) | 6 (7) | 2 (3) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 5 (5) | 3 (3) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.